CLINICAL TRIAL: NCT02719535
Title: Corneal Stiffness and Tangent Modulus to Predict the Rate of Corneal Curvature Change in Corneal Reshaping Therapy
Brief Title: Corneal Biomechanics and Corneal Reshaping Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B-Q46G
Record Dates: First submitted 2016-01-18; First posted 2016-03-25 (Estimated); Results first posted 2020-04-13 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2018-02

CONDITIONS: Myopia
Keywords: corneal reshaping therapy; corneal biomechanics
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Corneal reshaping therapy (Experimental): Subjects will be wearing corneal reshaping lenses for the correction of their myopia
  Interventions: Other: Corneal reshaping therapy

INTERVENTIONS:
Other: Corneal reshaping therapy — Reshaping the corneal curvature from wearing specific designed rigid gas permeable lenses

SUMMARY:
The aim of the proposed study is to investigate the predictive value of corneal biomechanical properties in corneal reshaping therapy and the role of these parameters in determining the amount of myopia reduction.

DETAILED DESCRIPTION:
Experiment 1: To evaluate changes in corneal biomechanics caused by short-term corneal reshaping therapy.

Subjects will wear a conventional RGP lens in one eye, randomly selected, and an orthokeratology lens in the fellow eye, for 30 minutes, 60 minutes and one night, respectively. Corneal stiffness and tangent modulus will be measured before and after each wearing period.

Experiment 2: To evaluate changes in and the recovery of corneal biomechanics effected by long-term corneal reshaping and to assess whether corneal biomechanics can predict the rate of corneal reshaping.

Subjects will wear orthokeratology lenses for 6 months. Regular follow up visits (1 week, 1 month, 3 months and 6 months) will be arranged to monitor the changes in corneal stiffness and tangent modulus.

ELIGIBILITY:
Inclusion Criteria:

* Myopia between -4D to -5D, with-the-rule astigmatism not more than 1.5D, spherical equivalent between -4D to -5.75D, difference between two eyes within 1D, best corrected spectacle visual acuity 0.10 logMAR in each eye

Exclusion Criteria:

* previous corneal reshaping therapy, long-term contact lens wear, ocular disease

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2016-01; Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew KC Lam, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Corneal Reshaping Therapy
Started | 59
Completed | 37
Not Completed | 22

BASELINE CHARACTERISTICS:
Groups:
- Corneal Reshaping Therapy: Participants receiving Corneal Reshaping Therapy were monitored for ocular biometry and refractive errors throughout a 6-month period. Corneal stiffness and tangent modulus were outcome measures.
Arm/Group | Corneal Reshaping Therapy
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 22 [18 to 30]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 37
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Hong Kong | 37

OUTCOME MEASURES:

1. Primary Outcome: Change of Corneal Stiffness From Baseline at 6 Months
Description: Corneal Stiffness: in N/mm Corneal parameters usually will stabilize in 1 month, this study will monitor it till 6 months.
Time Frame: At baseline, then change from baseline to 6 months
Measure: Mean (Standard Deviation); unit: N/mm
Groups:
- Treatment: Treatment
Arm/Group | Treatment
Number analyzed (Participants) | 37
N/mm | 0.061 (0.007)

2. Secondary Outcome: Change of Tangent Modulus From Baseline at 6 Months
Description: Tangent modulus: in MPa Corneal parameters usually will stabilize in 1 month, this study will monitor it till 6 months.
Time Frame: At baseline, then change from baseline to 6 months
Measure: Mean (Standard Deviation); unit: MPa
Arm/Group | Treatment
Number analyzed (Participants) | 37
MPa | 0.536 (0.118)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37
Other Adverse Events (participants affected / at risk) | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-25): https://cdn.clinicaltrials.gov/large-docs/35/NCT02719535/Prot_SAP_000.pdf